CLINICAL TRIAL: NCT00003202
Title: Alternating Phase I/II Trials of Twice-Weekly Infusion Gemcitabine (2'2'-Difluoro-2'-Deoxycytidine) and Concurrent Thoracic Radiation Alone - Or Following 2 Cycles of Cisplatin/Gemcitabine Induction Chemotherapy for the Treatment of Stage IIIA/IIIB Non Small Cell Lung Cancer (NSCLC)
Brief Title: Gemcitabine Plus Radiation Therapy or Combination Chemotherapy in Treating Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066052; CCCWFU-62197; NCI-G98-1386
Record Dates: First submitted 1999-11-01; First posted 2003-11-26 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Lung Cancer
Keywords: squamous cell lung cancer; large cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Cisplatin; Gemcitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase I/II trial to compare the effectiveness of gemcitabine with radiation therapy alone or following two-drug combination chemotherapy in treating patients with stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of twice-weekly gemcitabine when delivered concurrently with thoracic radiotherapy alone or following 2 cycles of induction chemotherapy in patients with Stage IIIA or IIIB non-small cell lung cancer.
* Assess the toxicity of concurrent thoracic radiation and gemcitabine in these patients.
* Determine the effectiveness of concurrent radiation and gemcitabine by determining the complete response rate, partial response rate, time to recurrence, pattern of recurrence, and overall survival in a cohort of these patients.

OUTLINE: This is an alternating two arm, dose escalation, multicenter study.

Arm I: Patients receive twice-weekly gemcitabine as a 30 minute infusion. Concurrent radiation therapy is administered 5 days a week for 6 weeks.

Arm II: Patients receive 2 cycles of induction chemotherapy consisting of gemcitabine as a 30 minute infusion on day 1 and 8 and cisplatin IV over 1 hour on day 1. Each cycle is 21 days. Patients then receive gemcitabine and radiation therapy as in arm I.

Cohorts of 3 patients are enrolled into each treatment arm at each dose level of gemcitabine. Toxicity for each arm is assessed independently. Once dose limiting toxicity (DLT) is observed at any dose level, 3 more patients are enrolled at the same dose level. The maximum tolerated dose (MTD) is defined as the dose at which no more than 1 of 6 patients experiences grade 4 toxicity, or no more than 4 of 6 patients experience grade 3 or worse toxicity (DLT). After the MTD is determined for each treatment arm, additional patients are treated at that dose level for the phase II portion of the study.

Patients are followed every 3 months for 2 years, then every 4 months for the next 2 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: There will be approximately 24-48 patients accrued into this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IIIA or IIIB non-small cell lung cancer that is unicentric and inoperable, including the following cellular types:

  * Squamous cell carcinoma
  * Adenocarcinoma
  * Bronchoalveolar carcinoma
  * Large cell anaplastic carcinoma
  * Non-small cell lung cancer not otherwise specified
* Tumors may be multifocal if all of disease is believed to be result of direct spread
* Disease must be fully accessible by radiotherapy ports for the entire prescribed dose
* No supraclavicular nodes or diffuse pleural involvement
* No contralateral hilar disease or an exudative, bloody, or cytologically malignant effusion
* Measurable disease required for phase II of this study

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* ECOG 0-2

Life expectancy:

* At least 1 year

Hematopoietic:

* Granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin greater than 10 g/dL

Hepatic:

* Bilirubin no greater than 2.0 mg/dL

Renal:

* BUN no greater than 1.5 times normal
* Creatinine no greater than 1.5 times normal

Pulmonary:

* FEV1 no greater than 1 liter except if tumor has negatively impacted
* pulmonary function

Other:

* No other serious medical or psychiatric illness
* No prior lung cancer except if free of disease for more than 3 years
* No other prior malignancy except nonmelanoma skin cancer or if free of
* disease for more than 1 year
* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior thoracic radiotherapy
* Concurrent radiotherapy to other anatomic sites allowed

Surgery:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1998-01; Primary Completion 2002-04 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
•Determine the maximum tolerated dose of twice-weekly gemcitabine when delivered concurrently with thoracic radiotherapy | 6 weeks

SECONDARY OUTCOMES:
assess the efficacy of dose of twice-weekly gemcitabine when delivered concurrently with thoracic radiotherapy | 72 days

CONTACTS AND LOCATIONS:
Overall Officials: Arthur William Blackstock, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina, United States